CLINICAL TRIAL: NCT02359175
Title: Supplementary Epidural Analgesia in Video-Assisted Thoracic Surgery (VATS) - The SEAVATS Study
Acronym: SEAVATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jimmy Højberg Holm, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13.034
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Lung Neoplasms; Pain; Immune Suppression
Keywords: Pain; Pain Measurement; VAS; Visual Analog Pain Scale; Analgesics; Opioid; Epidural analgesia; VATS; Video-assisted Thoracic Surgery; Lobectomy; Wedge Resection; Segmental Resection; Cytokins; Immune cells
MeSH Terms: conditions — Lung Neoplasms; Pain | interventions — Bupivacaine; Fentanyl; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Epidural analgesia (Active Comparator): Epidural catheter: Bupivacain 1,0 mg/ml + Fentanyl 2 micrograms/ml. Oral analgesia: Paracetamol, NSAID and placebo tablets.
  Interventions: Drug: Bupivacaine in epidural catheter; Drug: Fentanyl in epidural catheter; Drug: Oral Paracetamol; Drug: Oral NSAID; Drug: Placebo (for oral opioids)
- Placebo Epidural analgesia (Active Comparator): Epidural analgesia: Placebo. Oral analgesia: Paracetamol, NSAID and opioids tablets.
  Interventions: Drug: Placebo (for Bupivacain and Fentanyl i epidural catheter); Drug: Oral Paracetamol; Drug: Oral NSAID; Drug: Oral opioids

INTERVENTIONS:
Drug: Bupivacaine in epidural catheter — Bupivacain to be given in epidural catheter
  Arms: Active Epidural analgesia
Drug: Fentanyl in epidural catheter — Fentanyl to be given in epidural catheter
  Arms: Active Epidural analgesia
Drug: Placebo (for Bupivacain and Fentanyl i epidural catheter) — Saline to be given in epidural catheter
  Arms: Placebo Epidural analgesia
Drug: Oral Paracetamol — Paracetamol to be given orally
Drug: Oral NSAID — NSAID to be given orally
Drug: Oral opioids — Opioids to be given orally
  Arms: Placebo Epidural analgesia
Drug: Placebo (for oral opioids) — Placebo tablets to be given instead of oral opioids
  Arms: Active Epidural analgesia

SUMMARY:
Whereas it, in the case of conventional thoracotomy, has been demonstrated that thoracic epidural analgesia is more effective than systemic opioids in terms of pain relief and preservation of postoperative pulmonary function, the efficacy of epidural analgesia in video-assisted thoracic surgical (VATS) procedures, has not been sufficiently studied, but a beneficial effect might very well be present.

On the other hand, the risks associated with placement of a thoracic epidural catheter are well known and if similar pain relief can be achieved without it with no or only insignificant alternative side effects, this would be preferable.

The literature regarding the usefulness of epidural analgesia for reducing pain in Video-Assisted Thoracic Surgery is, at best, scarce with two small studies showing some effect and two showing no difference, none of the studies being blinded randomized controlled trials of adequate size.

The SEAVATS Study will try to answer this question.

DETAILED DESCRIPTION:
Study plan:

The hypothesis is that there is no difference in the amount of pain the patients will experience after VATS for pulmonary neoplasms.

Study design and setting:

The project is designed as a prospectively, double blinded, randomized, placebo controlled study comparing pain in two groups of patients.

Both groups of patients will:

* Have a epidural catheter placed.
* Receive a basis level of analgesics consisting of paracetamol and a nonsteroidal anti- inflammatory drug combined with a nerveblock placed intercostally during surgery.
* Have access to i.v. opioids as needed for any experienced pain after surgery.

One group of patients will be given local anaesthetics through the epidural catheter supplemented with placebo medication orally while the other group will receive saline in the epidural catheter supplemented with opioids orally.

Data collection:

Data will, during hospitalization, be collected in the operating theatre, in the postoperative care unit and in the surgical ward. Six months after surgery a questionnaire will be send to the patients to do follow-up regarding residual sequelae after surgery and placement of epidural catheter. Further follow-up with questionnaire has been planned for subsequent years.

As a secondary objective, in fifty-six of the patients from The SEAVATS Study, blood samples will be gathered during surgery and one hour and 24 hours after surgery, and compared with pre-operative levels.

These blood samples will be analysed for immune cells (NK-cells, levels and activity) and cytokines (IL-6, IL-10, IL-12 and IFN-gamma) as indicators of immunological response to surgery.

Research ethics:

The project has obtained ethics approval from The Regional Scientific Ethical Committees for Southern Denmark and acceptance to perform clinical research has been granted by The Danish Health and Medicines Authority. Consent to data collection has been provided by The Danish Data Protection Agency. Before entering the project, consent will be obtained from all patients. Rigorous data security will be maintained for five years and afterwards all data will be deleted. The Study is registered with The European Union Drug Regulating Authorities Clinical Trials Database (EudraCT) with EudraCT number 2014-000760-18 and is monitored by The Good Clinical Practice unit for Southern Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective VATS lobectomy, wedge- or segmental resection. (for the subsequent biomarker study, only lobectomy is a inclusion criteria, specified in protocol amendment July 27th 2016)
* Patient has accepted to have epidural analgesia as part of the anaesthesia for the procedure.
* Informed consent is attained.
* Patient is over 18 years of age.
* Patient is mentally able to answer questionnaires included in the study.

Exclusion Criteria:

* Allergies to any of the medications used in the trial.
* History of previous peptic ulcer.
* History of chronic pain to any degree that will interfere with quantification of pain postoperatively.
* Dementia or reduced mental capacity to any degree that will interfere with quantification of pain postoperatively.
* Pregnancy.
* Contra-indications to placement of epidural catheter.
* Any concurrent cancer disease or use of immune modulating drugs (criteria added as part of a protocol amendment July 27th 2016 for a subsequent biomarkers study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Intensity of pain (Self reported pain intensity) | 0-4 days
  Self reported pain intensity 5 times a day both in rest and during activity until chest tube is removed or day 4 after operation is reached.
Consumption "Rescue Analgesia" - i.v. opioids | 0-4 days
  The consumption of i.v. opioids is registered daily until chest tube is removed or day 4 after operation is reached.

SECONDARY OUTCOMES:
Duration of surgery | 0-4 days
  The duration of the surgical procedure will be registered.
Length of hospital stay | 0-4 days
  Admission time after surgery.
Time used placing epidural catheter | 0-4 days
  Procedural time and competence level of MD placing catheter
Side effects of epidural analgesia | 0-4 days
  Side effects observed using epidural analgesia including itching, nausea, vomiting, procedural pain, hypotension, dizziness, respiratory depression, reduced pulmonary function.
Sequelae following VATS and placement of epidural catheter | 60 months
  Questionnaire sent to patients 6, 12, 24 and 60 months after surgery. (criteria edited as part of a protocol amendment July 27th 2016 for a subsequent biomarkers study).

OTHER OUTCOMES:
Immune cells - NK cell levels. | During surgery and one hour and 24 hours after surgery, and compared with pre-operative levels.
  Levels of NK-cells will be examined as an indicator of immunological response to surgery.
  (The secondary outcomes "Immune cells", "Cytokines" and "Survival after VATS" should rightly have been registered in a separate sub study with a separate ClinicalTrials entry with "Immune cells - NK cell levels" as primary outcome measure and "Immune cells - NK cell activity", Cytokines" and "Survival after VATS" as a secondary outcomes as a separate sample size calculation was done to determine the needed inclusion for this part of the study. Now, instead, these outcomes will be defined as "Other Pre-specified Outcomes" with this explanation.)
Immune cells - NK cell activity. | During surgery and one hour and 24 hours after surgery, and compared with pre-operative levels.
  The NK-cell activity will be examined as an indicator of immunological response to surgery.
  (The secondary outcomes "Immune cells", "Cytokines" and "Survival after VATS" should rightly have been registered in a separate sub study with a separate ClinicalTrials entry with "Immune cells - NK cell levels" as primary outcome measure and "Immune cells - NK cell activity", Cytokines" and "Survival after VATS" as a secondary outcomes as a separate sample size calculation was done to determine the needed inclusion for this part of the study. Now, instead, these outcomes will be defined as "Other Pre-specified Outcomes" with this explanation.)
Cytokines | During surgery and one hour and 24 hours after surgery, and compared with pre-operative levels.
  Levels of cytokines (IL-6, IL-10, IL-12 and IFN-gamma) will be examined as indicators of immunological response to surgery.
  (The secondary outcomes "Immune cells", "Cytokines" and "Survival after VATS" should rightly have been registered in a separate sub study with a separate ClinicalTrials entry with "Immune cells - NK cell levels" as primary outcome measure and "Immune cells - NK cell activity", Cytokines" and "Survival after VATS" as a secondary outcomes as a separate sample size calculation was done to determine the needed inclusion for this part of the study. Now, instead, these outcomes will be defined as "Other Pre-specified Outcomes" with this explanation.)
Survival after VATS | 60 months
  Postoperative survival analysis. (The secondary outcomes "Immune cells", "Cytokines" and "Survival after VATS" should rightly have been registered in a separate sub study with a separate ClinicalTrials entry with "Immune cells" as primary outcome measure and "Cytokines" and "Survival after VATS" as a secondary outcomes as a separate sample size calculation was done to determine the needed inclusion for this part. Now, instead, these outcomes will be defined as "Other Pre-specified Outcomes" with this explanation.) (text initially added October 27th 2021, as the text was by mistake no included in the update after the protocol amendment 27 July 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy H Holm, MD, Principal Investigator — Department of Anaesthesia and Intensive Care - Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson J, Cheema S. Thoracic paravertebral nerve block. Br J Anaesth. 2006 Apr;96(4):537. doi: 10.1093/bja/ael038. No abstract available. PMID 16549628
- [Background] Kim JA, Kim TH, Yang M, Gwak MS, Kim GS, Kim MJ, Cho HS, Sim WS. Is intravenous patient controlled analgesia enough for pain control in patients who underwent thoracoscopy? J Korean Med Sci. 2009 Oct;24(5):930-5. doi: 10.3346/jkms.2009.24.5.930. Epub 2009 Sep 23. PMID 19794994
- [Background] Freise H, Van Aken HK. Risks and benefits of thoracic epidural anaesthesia. Br J Anaesth. 2011 Dec;107(6):859-68. doi: 10.1093/bja/aer339. Epub 2011 Nov 4. PMID 22058144
- [Background] Yie JC, Yang JT, Wu CY, Sun WZ, Cheng YJ. Patient-controlled analgesia (PCA) following video-assisted thoracoscopic lobectomy: comparison of epidural PCA and intravenous PCA. Acta Anaesthesiol Taiwan. 2012 Sep;50(3):92-5. doi: 10.1016/j.aat.2012.08.004. Epub 2012 Sep 7. PMID 23026166
- [Background] Yoshioka M, Mori T, Kobayashi H, Iwatani K, Yoshimoto K, Terasaki H, Nomori H. The efficacy of epidural analgesia after video-assisted thoracoscopic surgery: a randomized control study. Ann Thorac Cardiovasc Surg. 2006 Oct;12(5):313-8. PMID 17095972
- [Background] Fernandez MI, Martin-Ucar AE, Lee HD, West KJ, Wyatt R, Waller DA. Does a thoracic epidural confer any additional benefit following video-assisted thoracoscopic pleurectomy for primary spontaneous pneumothorax? Eur J Cardiothorac Surg. 2005 Apr;27(4):671-4. doi: 10.1016/j.ejcts.2004.12.045. PMID 15784372
- [Derived] Holm JH, Andersen C, Licht PB, Toft P, Zegers FD, Lambertsen KL, Brochner AC. Immunological effects of post-operative epidural analgesia versus oral opioids in VATS. Dan Med J. 2024 Sep 9;71(10):A09230582. doi: 10.61409/A09230582. PMID 39323258
- [Derived] Holm JH, Andersen C, Toft P. Epidural analgesia versus oral morphine for postoperative pain management following video-assisted thoracic surgery: A randomised, controlled, double-blind trial. Eur J Anaesthesiol. 2024 Jan 1;41(1):61-69. doi: 10.1097/EJA.0000000000001921. Epub 2023 Nov 15. PMID 37962202